CLINICAL TRIAL: NCT04594343
Title: A Randomized, Double-blind, Placebo-controlled Safety and Clinical Outcomes Study of Disulfiram in Subjects With Moderate COVID-19
Brief Title: Clinical Study to Evaluate the Effects of Disulfiram in Patients With Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETICA (Other)
Collaborators: Spring Research Foundation (Network)
Responsible Party: Principal Investigator, Augusto Mota, Principal Investigator, ETICA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR-001-201
Record Dates: First submitted 2020-10-18; First posted 2020-10-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Disulfiram

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either the active product (disulfiram) or placebo.
  Disulfiram will be dosed 500 mg daily for a total of 14 days of treatment. A matching placebo will be given using the same dosing schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In order to minimize bias due to key baseline characteristics that can impact clinical outcomes, the randomization will be stratified 1:1 to placebo or active product based on age and comorbidities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Disulfiram (Experimental)
  Interventions: Drug: Disulfiram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Disulfiram — The subject will receive 500 mg of disulfiram orally or enterally through NG tube if in mechanical ventilation once daily for 14 days
  Other Names: Antabuse
  Arms: Disulfiram
Drug: Placebo — The subject will receive a matching placebo orally or enterally through NG tube if in mechanical ventilation once daily for 14 days
  Arms: Placebo

SUMMARY:
This clinical trial evaluates the safety, efficacy, and biomarker levels of FDA-approved drug disulfiram in the treatment of adult subjects hospitalized with moderate COVID-19. Disulfiram may limit the hyperinflammatory response associated with COVID-19 and reduce the risk of progression to severe illness.

Subjects will be screened and randomized to receive either daily administration of oral disulfiram or placebo for 14 days. Subjects will be followed up on Day 28.

DETAILED DESCRIPTION:
COVID-19 is a respiratory disease caused by a novel coronavirus (SARS-CoV-2) and causes substantial morbidity and mortality. There is currently no vaccine to prevent COVID-19 or infection with SARS-CoV-2 or therapeutic agent to treat COVID-19. The ongoing COVID-19 pandemic has demonstrated increased risk to those with an aging immune system. The elderly and those with comorbidities are reported as being the most susceptible to COVID-19, which may be due to a higher basal state of inflammation ("inflammaging") and a primed inflammasome pathway. Disulfiram, an FDA-approved drug for the treatment of alcohol dependence, has a potential for limiting the hyperinflammatory response associated with COVID-19. Specifically, the drug inhibits gasdermin D pore formation, reducing pyroptosis and netosis and could target the root cause of hyperinflammation, weakening the cytokine storm and therefore reducing the risk of progression to severe illness.

This is a stratified, randomized, double-blind, placebo-controlled study of disulfiram in hospitalized subjects over the age of 50 diagnosed with moderate COVID-19. Up to 200 subjects are planned to be enrolled and randomized (1:1) to either receive 500 mg of disulfiram (active product) or placebo, orally (po) or enterally (only in patients that require mechanical ventilation) once daily for fourteen (14) days in addition to standard of care. Stratification will be done at randomization based on age and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled in the study only if all the inclusion criteria are met.

1. Male and female subjects, age 35 or older.
2. Female subjects of childbearing potential must have a negative hCG (in urine or blood) pregnancy test.
3. An International Ethics Committee (IEC) approved informed consent is signed and dated prior to any study-related activities.
4. Willing to abstain from any alcohol or substances containing alcohol (including medications, personal hygiene products, salad dressing) within 24 hours prior to treatment and for 14 days after treatment concludes.
5. Have the ability to understand the requirements of the study and is willing to comply with all study procedures and visits.
6. Respiratory rate: ≤ 30 per minute.
7. Use supplemental O2 via nasal cannula or equivalent.
8. Currently hospitalized ≤ 5 days.
9. PCR test or rapid antigen test confirming SARS-CoV-2.
10. In the opinion of the investigator, able to participate in the study.

Exclusion Criteria:

Subjects may not be enrolled in the study if any of the exclusion criteria apply.

1. Admission into the Intensive Care Unit (ICU) at screening and baseline.
2. Clinically active Hepatitis.
3. ALT or AST > 3 times the upper limit of normal.
4. Need for invasive or non-invasive ventilation at screening and baseline.
5. Stage 4 severe chronic kidney disease or requiring dialysis or estimated GFR < 30.
6. Known allergy to disulfiram.
7. Treatment with any of the medications listed below within 7 days prior to the baseline visit 1: Amprenavir, Dronabinol, Hydantoins, Metronidazole, Ritonavir, Benznidazole, Dyphylline, Idelalisib, Naltrexone, Sertraline, Chloral Hydrate, Ethanol, Immuno-modulatory drugs, Paclitaxel, Tinidazole, Cocaine, Ethotoin, Ixabepilone, Phenytoin, Tipranavir, Cyclosporine, Fosphenytoin, Lithium, Pimozide, Tranylcypromine, Dasabuvir, Guaifenesin, Mesoridazine, Pirfenidone.
8. Participation in any other interventional trial within 30 days prior to enrollment.
9. Active malignancy (excluding basal cell carcinoma, squamous cell carcinoma, in situ cervical cancer, or adenocarcinoma of the prostate with low or very low-risk categories by NCCN criteria).
10. Any surgical or medical condition which in the opinion of the investigator may interfere with participation in the study or which may affect the outcome of the study.
11. Fully vaccinated for COVID-19 (number of doses as per manufacturer recommendation.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | From enrollment to clinical improvement (1 point or more in the WHO score), up to 28 days
  Defined as the time from baseline to the first post-baseline assessment with an improvement in WHO score of ≥1 point.

SECONDARY OUTCOMES:
Mean number of days of supplemental oxygen (WHO score ≥4) | Baseline to Day 28
Time to discharge from the hospital | From baseline to discharge, up to 28 days.
Percentage of subjects that are discharged by Day 8 | At Day 8
Percentage of subjects that worsened 1 or more points on the WHO Ordinal Scale, from baseline to any post baseline assessment through Day 28. | Baseline to Day 28
Mean number of days of non-invasive ventilation or high flow oxygen devices or invasive mechanical ventilation (WHO Score 5 or 6) over the 28-day period. | Baseline to Day 28
Mean number of days subjects were in the Intensive Care Unit (ICU) | Baseline to Day 28
Percentage of subjects that were on non-invasive ventilation or high flow oxygen devices or invasive mechanical ventilation (WHO Score 5 or 6) over the 28-day period. | Baseline to Day 28
28-day mortality | At Day 28

OTHER OUTCOMES:
Change from baseline to Day 8 and Day 15 for cytokine IL-18 | Baseline, Day 8 and Day 15
  Mean change and percent change
Percentage of subjects requiring supplemental oxygen (WHO Score ≥4) by Day 8, 15, and 28. | Baseline, Day 8, Day 15 and Day 28
Percentage of subjects that are discharged by Day 15 and Day 28. | Day 15 and Day 28
Percentage of subjects that worsened 1 or more points on the WHO Ordinal Scale from baseline through Day 8 and Day 15. | Baseline to Day 8, 15
Percentage of subjects admitted to the Intensive Care Unit. | Baseline to Day 28
Percentage of subjects that improved 1 or more points on the WHO Ordinal Scale from baseline to Day 8, 15, and 28. | Baseline to Day 8, 15, and 28
Change in total neutrophil count from baseline to Day 8 and 15. | Baseline, Day 8 and Day 15
  Mean change and percent change
Percent change in total lymphocyte count from baseline to Day 8 and Day 15 | Baseline, Day 8 and Day 15
Change from baseline to Day 8 and Day 15 for neutrophil-derived circulating free DNA (cf-DNA/NETs) | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for Cytokine TNF-α | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for cytokine IL-1β | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for cytokine IL-1RA | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for cytokine IL-6 | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for cytokine IL-8 | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for cytokine IL-10 | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for Lactate Dehydrogenase (LDH) | Baseline, Day 8 and Day 15
  Mean change and percent change
Change from baseline to Day 8 and Day 15 for D-dimer | Baseline, Day 8 and Day 15
  Mean change and percent change
Association between baseline and worst post-baseline WHO score | Baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Mota, MD/PhD, Principal Investigator — ETICA; Wendy Cousin, PhD, Study Director — Spring Research Foundation
Locations (1):
- ETICA, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Saifi MA, Shaikh AS, Kaki VR, Godugu C. Disulfiram prevents collagen crosslinking and inhibits renal fibrosis by inhibiting lysyl oxidase enzymes. J Cell Physiol. 2022 May;237(5):2516-2527. doi: 10.1002/jcp.30717. Epub 2022 Mar 13. PMID 35285015